CLINICAL TRIAL: NCT04442672
Title: The Value of Multimodal Monitoring in the Treatment of Compartment Syndrome: a Study Based on Healthy Volunteers
Brief Title: Early Diagnosis of Compartment Syndrome by Multimodal Detection Technique
Acronym: MMCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: I2019001099
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2019-07

CONDITIONS: Compartment Syndrome of Leg
Keywords: compartment syndromes; multimodal; Ultrasonography; Near-Infrared Spectroscopy
MeSH Terms: conditions — Compartment Syndromes | interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- compartment syndrome model group(CSM group) (Experimental)
  Interventions: Procedure: acute compartment syndrome model of health volunteer
- sham group (Sham Comparator)
  Interventions: Procedure: sham

INTERVENTIONS:
Procedure: acute compartment syndrome model of health volunteer — the acute compartment syndrome model of health volunteer is induced by pressurizing the calves by the cuff, and the cuff is inflated and pressurized to a pressure value of 20, 30, 40, 50, 60, 70, 80 mmHg. the pressure inside the cuff was up to 10 s during pressurization and maintained stable for 1 min, measured and the above indicators were recorded within 3 min.
  Arms: compartment syndrome model group(CSM group)
Procedure: sham — surrounding the cuff but not inflate it.
  Arms: sham group

SUMMARY:
compartment syndrome has a high incidence in patients with a variety of diseases, including fractures, and delayed diagnosis or without intervention can lead to severe adverse prognosis, such as limb deformities, amputations and even death. Early diagnosis and early intervention are important, especially early diagnosis. Now, the diagnosis of compartment syndrome in clinical is based on medical history, clinical manifestations and measuring the compartment pressure by fine needle puncture. However, this diagnostic method is not easy to achieve early accurate diagnosis and non-invasive continuous monitoring. The study found that the increase of compartment pressure can lead to local changes of hemodynamic, tissue metabolism and nerve function. There are also studies and reports of near-infrared spectral tissue oxygen measurement technology, ultrasonic Doppler technology, near-infrared spectral pulse oxygen measurement technology and infrared thermal imaging technology can be used for noninvasive monitoring of acute compartment syndrome, but it is not clear that which is better above in early diagnosis of acute compartment syndrome.

The purpose of this study was to simulate the process of early pressure increase in the compartment by pressurizing the volunteers' calves by cuff, and then measured the tissue oxygen in the Anterior fascia compartment using a non-invasive monitor of the tissue oxygen parameters, the ultrasonic machine measured the blood flow signal of the upper and lower backbone blood vessels, and the blood oxygen meter to measure the blood saturation of the upper and lower ends of the limb. The infrared thermal imager measured the near and far limb temperature of the hemostatic belt and the two-point identification of the skin sensory nerve function at the far end of the fascia chamber. Then compare the correlation of these indicators with pressure changes.

DETAILED DESCRIPTION:
The participants is health volunteers, age 18-60 years. When the participants agree to participate in the experiment, the experimenter first needs to explain the experimental process to the participants, and ask the participants to agree and sign the informed consent before they can conduct the experiment. The experiment was conducted in the emergency medicine department of a university-affiliated top three hospital.

When the participants are included in the experimental study, the general demographic information of the participants, such as name, gender, age, etc., is first collected. Ensure the experimental environment is comfortable, ambient temperature 20-24℃, ambient humidity 50-60%. Participants have loose clothing on their lower limbs to avoid pressure on their limbs. Take the supine position, keep the calf hanging, support the heel, make the calf level flush with the heart, rest for 5 minutes.

The monitor (M3002A, Philips Medizin Systeme Boeblingen GmbH, Germany) was used to continuously monitor the electrocardiogram, the left upper arm measured blood pressure (BP), and the right middle finger to monitor pulse oximetry (SpO2). The calf circumference was measured at the midpoint of the bilateral humerus with a soft ruler. The maximum thickness of anterior fascia compartment was measured at the midpoint of the tibia using an ultrasonic machine (Acclarix AX8, Shenzhen Libang Precision Instrument Co., Ltd., China).

The random number table method selects one side of the calf as the experimental side and the opposite side as the control side.

(8) The following parameters were recorded at baseline (pressure 0mmHg in the calf tourniquet on both sides): (1) heart rate, blood pressure; (2) right middle finger, lower limbs, middle toe finger vein oxygen SpO2; (3) bilateral Local blood tissue parameters (TOI, THI, ΔCHb, CHbO2, ΔCtHb) in the calf; (4) Near-infrared thermography temperature values (T-u1, T-u2) in the knee and thighs of the lower leg and the instep and toe Near-infrared thermography temperature values (T-d1, T-d2); (5) bilateral radial artery ultrasound Doppler measurement parameters (D-pa, S-pa, Vs-pa, Vd-pa, DRAF-pa) Ultrasound Doppler measurement parameters of bilateral iliac veins (D-pv, S-pv, Vs-pv, Vd-pv), bilateral posterior tibial artery and dorsal artery ultrasound Doppler measurement parameters (Vs-pta, Vd -pta, SFAF-pta, Vs-da, Vd-da, SFAF-da). (6) Two-point identification threshold TPD.

In turn, the experimental side calf tourniquet was inflated and pressurized to a pressure value of 20, 30, 40, 50, 60, 70, 80 mmHg, and the pressure inside the tourniquet was up to 10 s during pressurization, and maintained stable for 1 min, measured and the above indicators were recorded within 3 min. During the experiment, the subjects were closely monitored for adverse reactions. At the end of the study, the observation was continued for 30 minutes, and the drinking water was at least 500 ml, and the limb sensation, pain and urine color were continuously observed within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, aged 18-60 years; No obvious cardiovascular diseases such as cardiovascular and cerebrovascular diseases; Complete limbs without deformity and no history of lower limb trauma; Informed consent

Exclusion Criteria:

* pregnancy or use of oral contraceptives; History of diabetes; History of deep vein thrombosis; Peripheral neuropathy; peripheral vascular disease; History of rhabdomyolysis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Blood flow spectrum of the radial artery and dorsal artery by ultrasound Doppler examination | 40 minutes
  During the cuff compression, the blood flow spectrum of the radial artery and dorsal artery was recorded by the ultrasound, and analyzed later for the blood direction and duration.
tissue oxygen of the compartment by Infrared oxygen saturation monitor | 40 minutes
  The infrared oxygen saturation monitor probe is placed on the anterior surface of the anterior fascia, and the changes of tissue oxygen index are continuously monitored during the process of cuff compression.

SECONDARY OUTCOMES:
temperture changes by near-infrared thermography | 40min
  The temperature of the proximal and distal skin of the fascial compartment is continuously monitored by near-infrared thermography
Pulse oxygen | 40 minutes
  the pulse oxygen of right middle finger, lower limbs, middle toe finger is continuously monitored
Systemic hemodynamics | 40 minutes
  heart rate, blood pressure is continuously monitored
Two-point identification check | 40 minutes
  Two-point identification check of the back of foot is monitored during each pressure level

CONTACTS AND LOCATIONS:
Overall Officials: Mao Zhang, PHD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, Zhejiang University School of Medicine Institute of Emergency Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shadgan B, Pereira G, Menon M, Jafari S, Darlene Reid W, O'Brien PJ. Risk factors for acute compartment syndrome of the leg associated with tibial diaphyseal fractures in adults. J Orthop Traumatol. 2015 Sep;16(3):185-92. doi: 10.1007/s10195-014-0330-y. Epub 2014 Dec 28. PMID 25543232
- [Background] Olson SA, Glasgow RR. Acute compartment syndrome in lower extremity musculoskeletal trauma. J Am Acad Orthop Surg. 2005 Nov;13(7):436-44. doi: 10.5435/00124635-200511000-00003. PMID 16272268
- [Background] McQueen MM, Duckworth AD. The diagnosis of acute compartment syndrome: a review. Eur J Trauma Emerg Surg. 2014 Oct;40(5):521-8. doi: 10.1007/s00068-014-0414-7. Epub 2014 Jun 3. PMID 26814506
- [Background] Mubarak SJ, Hargens AR. Acute compartment syndromes. Surg Clin North Am. 1983 Jun;63(3):539-65. doi: 10.1016/s0039-6109(16)43030-6. No abstract available. PMID 6346542
- [Background] von Keudell AG, Weaver MJ, Appleton PT, Bae DS, Dyer GSM, Heng M, Jupiter JB, Vrahas MS. Diagnosis and treatment of acute extremity compartment syndrome. Lancet. 2015 Sep 26;386(10000):1299-1310. doi: 10.1016/S0140-6736(15)00277-9. PMID 26460664
- [Background] Shadgan B, Menon M, Sanders D, Berry G, Martin C Jr, Duffy P, Stephen D, O'Brien PJ. Current thinking about acute compartment syndrome of the lower extremity. Can J Surg. 2010 Oct;53(5):329-34. PMID 20858378
- [Background] Soller BR, Yang Y, Soyemi OO, Ryan KL, Rickards CA, Walz JM, Heard SO, Convertino VA. Noninvasively determined muscle oxygen saturation is an early indicator of central hypovolemia in humans. J Appl Physiol (1985). 2008 Feb;104(2):475-81. doi: 10.1152/japplphysiol.00600.2007. Epub 2007 Nov 15. PMID 18006869
- [Result] Mancini DM, Bolinger L, Li H, Kendrick K, Chance B, Wilson JR. Validation of near-infrared spectroscopy in humans. J Appl Physiol (1985). 1994 Dec;77(6):2740-7. doi: 10.1152/jappl.1994.77.6.2740. PMID 7896615
- [Result] Shuler MS, Reisman WM, Kinsey TL, Whitesides TE Jr, Hammerberg EM, Davila MG, Moore TJ. Correlation between muscle oxygenation and compartment pressures in acute compartment syndrome of the leg. J Bone Joint Surg Am. 2010 Apr;92(4):863-70. doi: 10.2106/JBJS.I.00816. PMID 20360509
- [Result] Breit GA, Gross JH, Watenpaugh DE, Chance B, Hargens AR. Near-infrared spectroscopy for monitoring of tissue oxygenation of exercising skeletal muscle in a chronic compartment syndrome model. J Bone Joint Surg Am. 1997 Jun;79(6):838-43. doi: 10.2106/00004623-199706000-00006. PMID 9199380
- [Result] Cathcart CC, Shuler MS, Freedman BA, Reno LR, Budsberg SC. Correlation of near-infrared spectroscopy and direct pressure monitoring in an acute porcine compartmental syndrome model. J Orthop Trauma. 2014 Jun;28(6):365-9. doi: 10.1097/BOT.0b013e3182a75ceb. PMID 24857905
- [Result] Gentilello LM, Sanzone A, Wang L, Liu PY, Robinson L. Near-infrared spectroscopy versus compartment pressure for the diagnosis of lower extremity compartmental syndrome using electromyography-determined measurements of neuromuscular function. J Trauma. 2001 Jul;51(1):1-8, discussion 8-9. doi: 10.1097/00005373-200107000-00001. PMID 11468459
- [Result] Arbabi S, Brundage SI, Gentilello LM. Near-infrared spectroscopy: a potential method for continuous, transcutaneous monitoring for compartmental syndrome in critically injured patients. J Trauma. 1999 Nov;47(5):829-33. doi: 10.1097/00005373-199911000-00002. PMID 10568708
- [Result] Schmidt AH, Bosse MJ, Obremskey WT, O'Toole RV, Carroll EA, Stinner DJ, Hak DJ, Karunakar M, Hayda R, Frey KP, Di J, Zipunnikov V, MacKenzie E; Major Extremity Trauma Research Consortium (METRC). Continuous Near-Infrared Spectroscopy Demonstrates Limitations in Monitoring the Development of Acute Compartment Syndrome in Patients with Leg Injuries. J Bone Joint Surg Am. 2018 Oct 3;100(19):1645-1652. doi: 10.2106/JBJS.17.01495. PMID 30277994
- [Result] Garr JL, Gentilello LM, Cole PA, Mock CN, Matsen FA 3rd. Monitoring for compartmental syndrome using near-infrared spectroscopy: a noninvasive, continuous, transcutaneous monitoring technique. J Trauma. 1999 Apr;46(4):613-6; discussion 617-8. doi: 10.1097/00005373-199904000-00009. PMID 10217223
- [Result] Lima A, Bakker J. Near-infrared spectroscopy for monitoring peripheral tissue perfusion in critically ill patients. Rev Bras Ter Intensiva. 2011 Sep;23(3):341-51. English, Portuguese. PMID 23949407
- [Result] Boezeman RP, Becx BP, van den Heuvel DA, Unlu C, Vos JA, de Vries JP. Monitoring of Foot Oxygenation with Near-infrared Spectroscopy in Patients with Critical Limb Ischemia Undergoing Percutaneous Transluminal Angioplasty: A Pilot Study. Eur J Vasc Endovasc Surg. 2016 Nov;52(5):650-656. doi: 10.1016/j.ejvs.2016.07.020. Epub 2016 Sep 7. PMID 27614555
- [Result] Feldman F, Nickoloff EL. Normal thermographic standards for the cervical spine and upper extremities. Skeletal Radiol. 1984;12(4):235-49. doi: 10.1007/BF00349505. PMID 6505731
- [Result] Uematsu S, Edwin DH, Jankel WR, Kozikowski J, Trattner M. Quantification of thermal asymmetry. Part 1: Normal values and reproducibility. J Neurosurg. 1988 Oct;69(4):552-5. doi: 10.3171/jns.1988.69.4.0552. PMID 3418388
- [Result] Thangam S, Vaz M, Kurpad AV, Shetty PS. Superficial thermal gradients during mild body cooling and its relationship to forearm blood flow. Indian J Physiol Pharmacol. 1993 Oct;37(4):328-32. PMID 8112811
- [Result] Katz LM, Nauriyal V, Nagaraj S, Finch A, Pearlstein K, Szymanowski A, Sproule C, Rich PB, Guenther BD, Pearlstein RD. Infrared imaging of trauma patients for detection of acute compartment syndrome of the leg. Crit Care Med. 2008 Jun;36(6):1756-61. doi: 10.1097/CCM.0b013e318174d800. PMID 18496371
- [Result] Theuma F, Cassar K. The use of smartphone-attached thermography camera in diagnosis of acute lower limb ischemia. J Vasc Surg. 2018 Apr;67(4):1297. doi: 10.1016/j.jvs.2017.02.054. No abstract available. PMID 29579472
- [Result] Lin PH, Saines M. Assessment of lower extremity ischemia using smartphone thermographic imaging. J Vasc Surg Cases Innov Tech. 2017 Oct 14;3(4):205-208. doi: 10.1016/j.jvscit.2016.10.012. eCollection 2017 Dec. PMID 29349425
- [Result] Turnipseed WD, Hurschler C, Vanderby R Jr. The effects of elevated compartment pressure on tibial arteriovenous flow and relationship of mechanical and biochemical characteristics of fascia to genesis of chronic anterior compartment syndrome. J Vasc Surg. 1995 May;21(5):810-6; discussion 816-7. doi: 10.1016/s0741-5214(05)80012-6. PMID 7769739
- [Result] Wiebe S, Kellenberger CJ, Khoury A, Miller SF. Early Doppler changes in a renal transplant patient secondary to abdominal compartment syndrome. Pediatr Radiol. 2004 May;34(5):432-4. doi: 10.1007/s00247-003-1094-3. Epub 2003 Dec 17. PMID 14685790
- [Result] Kirkpatrick AW, Colistro R, Laupland KB, Fox DL, Konkin DE, Kock V, Mayo JR, Nicolaou S. Renal arterial resistive index response to intraabdominal hypertension in a porcine model. Crit Care Med. 2007 Jan;35(1):207-13. doi: 10.1097/01.CCM.0000249824.48222.B7. PMID 17080005
- [Result] Auerbach DN, Bowen AD 3rd. Sonography of leg in posterior compartment syndrome. AJR Am J Roentgenol. 1981 Feb;136(2):407-8. doi: 10.2214/ajr.136.2.407. No abstract available. PMID 6781266
- [Result] Mc Loughlin S, Mc Loughlin MJ, Mateu F. Pulsed Doppler in simulated compartment syndrome: a pilot study to record hemodynamic compromise. Ochsner J. 2013 Winter;13(4):500-6. PMID 24357997
- [Result] Rosales-Velderrain A, Padilla M, Choe CH, Hargens AR. Increased microvascular flow and foot sensation with mild continuous external compression. Physiol Rep. 2013 Dec 19;1(7):e00157. doi: 10.1002/phy2.157. eCollection 2013 Dec 1. PMID 24744851
- [Result] Clayton JM, Hayes AC, Barnes RW. Tissue pressure and perfusion in the compartment syndrome. J Surg Res. 1977 Apr;22(4):333-9. doi: 10.1016/0022-4804(77)90152-4. No abstract available. PMID 850397
- [Result] Lynch JE, Lynch JK, Cole SL, Carter JA, Hargens AR. Noninvasive monitoring of elevated intramuscular pressure in a model compartment syndrome via quantitative fascial motion. J Orthop Res. 2009 Apr;27(4):489-94. doi: 10.1002/jor.20778. PMID 18979529